CLINICAL TRIAL: NCT05475054
Title: Indications, Trends, and Perioperative Outcomes of Minimally Invasive and Open Liver Surgery in Non-obese and Obese Patients: an International Multicentre Propensity Score Matched Retrospective Cohort Study of 9963 Patients.
Brief Title: Impact of Minimally Invasive and Open Liver Surgery in Different BMI-classes
Acronym: MILSOBES
Status: Completed | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); The Queen Elizabeth Hospital (Other); Umberto I Mauriziano Hospital, Turin, Italy (Unknown); Oslo University Hospital and Institute of Medicine, University of Oslo, Oslo, Norway (Unknown); Padua University Hospital, Padua, Italy (Unknown); IRCCS San Raffaele (Other); University Hospital of Girona Dr. Josep Trueta (Network); Clinica Universidad de Navarra, Pamplona, Spain (Unknown); Institut Mutualiste Montsouris, Université Paris Descartes, Paris, France (Unknown); Groeninge Hospital, Kortrijk, Belgium (Unknown); University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom (Unknown); Riuniti Hospital, Polytechnic University of Marche, Ancona, Italy (Unknown); University of Verona, Verona, Italy (Unknown); Virginia Mason Medical Center, Seattle, USA (Unknown); University of California San Francisco, California, USA (Unknown); Moscow Clinical Research Centre, Moscow, Russia (Unknown); Università Cattolica del Sacro Cuore-IRCCS, Rome, Italy (Unknown); Antoine Béclère Hospital, Paris, France (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor
Other Study IDs: NP5469
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Liver Cancer; Liver Metastases; Obesity
Keywords: overweight; fatty liver; open liver resection; laparoscopic liver resection; minimally invasive liver resection
MeSH Terms: conditions — Liver Neoplasms; Obesity; Overweight; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open liver resection: Non-obese or obese patients that underwent an open liver resection for all indications
- Minimally invasive liver resection: Non-obese or obese patients that underwent a minimally invasive liver resection for all indications
  Interventions: Procedure: Minimally invasive liver resection

INTERVENTIONS:
Procedure: Minimally invasive liver resection — A liver resection performed by minimally invasive (keyhole) surgery
  Other Names: Laparoscopic liver resection
  Groups: Minimally invasive liver resection

SUMMARY:
Despite the worldwide increase of both obesity and use of minimally invasive liver surgery(MILS), evidence regarding the safety and eventual benefits of MILS in obese patients is scarce. The aim of this study is therefore to compare the outcomes of non-obese and obese patients(BMI 18.5-29.9 and BMI≥30, respectively) undergoing MILS and OLS, and to assess trends in MILS use among obese patients. In this retrospective cohort study, patients operated at 20 hospitals in eight countries(2009-2019) will be included and the characteristics and outcomes of non-obese and obese patients will be compared. Thereafter, the outcomes of MILS and OLS were compared in both groups after propensity-score matching(PSM). Changes in the adoption of MILS during the study period will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients that have undergone an elective minimally invasive or open liver resection

Exclusion Criteria:

* Patients that have undergone a hand-assisted or robotic procedure
* Patients with a BMI lower than 18.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent an elective liver resection at 20 hepatobiliary referral centres between January 2009 and December 2019
Sampling Method: Non-Probability Sample
Enrollment: 9963 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Major complications | 30 days postoperatively
  Severe complications (Clavien-Dindo grade 3a or higher) related to the surgical procedure

SECONDARY OUTCOMES:
Overall complications | 30 days postoperatively
  Overall complications related to the surgical procedure
Length of hospital stay | 30 days postoperatively
  The length of hospital stay for the surgical procedure
R0 resection margin | 30 days postoperatively
  Proportion of patients in whom a microscopically radical resection of both the primary colorectal carcinoma and the liver metastases was performed.
  Proportion of patients in whom a microscopically radical resection was performed
Intraoperative blood loss | During the surgical procedure
  Intraoperative blood loss in milliliters
Operative time | During the surgical procedure
  Operative time in minutes
Conversion to open surgery | During the surgical procedure
  Intra-operative conversion to an open or hand-assisted procedure in the minimally invasive group
Respiratory complications | 30 days postoperatively
  All respiratory complications
Wound-related complications | 30 days postoperatively
  All wound-related complications
Post-hepatectomy liver failure | 30 days postoperatively
  Occurrence of post-hepatectomy liver failure (ISGLS definition and classification)
Bile leak | 30 days postoperatively
  Occurrence of bile leak (ISGLS definition and classification)
Ascites | 30 days postoperatively
  Occurrence of ascites
Mortality | 90 days postoperatively
  Postoperative mortality
Red blood cell transfusion | During the surgical procedure
  Intraoperative red blood cell transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The data of this study will be available from the corresponding author, Professor Mohammed Abu Hilal, upon reasonable request. The data are not publicly available since this could compromise the privacy of research participants.